CLINICAL TRIAL: NCT06498154
Title: Eliminating Breast Surgery for Triple Negative or HR-/HER2+ Breast Cancer Patients With Clinical Complete Response to Combined Neoadjuvant Chemotherapy and Neoadjuvant Radiotherapy: A Multicenter, Phase 2 Trial (EBCS)
Brief Title: Eliminating Breast Surgery for Breast Cancer Patients With Clinical Complete Response to Neoadjuvant Systemic Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other); The First Affiliated Hospital of Hainan Medical University (Other Government); Shandong Cancer Hospital and Institute (Other); First Affiliated Hospital of Kunming Medical University (Other); Chongqing University Cancer Hospital (Other); Tangshan People's Hospital (Other); Taizhou Hospital (Other)
Responsible Party: Principal Investigator, Xuchen Cao, MD, Tianjin Medical University Cancer Institute and Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TianJin Medical University....
Record Dates: First submitted 2024-07-06; First posted 2024-07-12 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Intervention Model Description: Chemotherapy combined with radiotherapy
Masking Description: Masking Description
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant Chemotherapy combined with Neoadjuvant Radiotherapy (Experimental): Patients who meet the criteria for enrollment initially receive four cycles of TCb (HP) * neoadjuvant chemotherapy, followed by neoadjuvant radiotherapy starting from the fifth cycle of TCb (HP) * neoadjuvant chemotherapy. After completion of six cycles of neoadjuvant chemotherapy, patients underwent breast magnetic resonance imaging. When a patient meets the MRI criteria suggestive of a complete clinical response (cCR), vacuum assisted core biopsy (VACB) targeting the primary lesion is performed under ultrasound or stereotactic guidance. A minimum of six cores, are obtained using a 7-10 G needle. Biopsy specimens are examined by a pathologist to assess the residual tumor and tumor bed. When no tumor or atypical cells are confirmed in the valid VACB specimen, breast and axillary surgery will be omitted.
  Interventions: Radiation: Neoadjuvant Chemotherapy combined with Neoadjuvant Radiotherapy

INTERVENTIONS:
Radiation: Neoadjuvant Chemotherapy combined with Neoadjuvant Radiotherapy — Neoadjuvant radiotherapy: whole-breast irradiation ( 50 Gy in 25 fractions) plus a mandatory boost (14 Gy in seven fractions, which began on the day following completion of whole-breast irradiation) TCb (HP) * : Triple negative patients will receive TCb regimens with or without immunotherapy and HER2 positive patients will receive TCb(HP) regimens.

SUMMARY:
Phase II multicenter prospective study on the safety of eliminating surgery for triple negative or HER2 positive breast cancer patients with clinical response to neoadjuvant radiotherapy and neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
The main purpose: To explore the safety of eliminating surgery for triple negative or HER2 positive breast cancer patients with clinical response to neoadjuvant chemoradiotherapy. Secondary study objective: To explore predictive molecular biomarkers of response to neoadjuvant chemoradiotherapy and investigate whether ctDNA can predict pCR or survival outcome.

Primary endpoint: 5-year event-free survival (5-year EFS). Secondary end points: Whether combined neoadjuvant chemoradiotherapy can improve breast pathological complete response rate (bpCR: ypT0), overall survival (OS), patient-reported outcomes (PROs) and safety

ELIGIBILITY:
Inclusion Criteria:

* Female initial treatment patients aged ≥ 18 years and ≤ 70 years old
* ECOG score 0-1
* Clinical T1-2N0 HER2 positive ( HR negative HER2 IHC score of 3+, or 2+and ISH test positive) or triple negative invasive breast cancer
* Left ventricular ejection fraction (LVEF) ≥ 50%
* 12 lead electrocardiogram: QT interval (QTcF) corrected by Fridericia method for females<470ms
* The functional level of the main organs must meet the following requirements: blood routine: ANC ≥ 1.5 × 109/L# PLT≥90 × 109/L# Hb≥90 g/L#Blood biochemistry: TBIL ≤ 2.5 × ULN# ALT and AST ≤ 2.5 × ULN# BUN and Cr ≤ 1.5 × ULN#
* For female subjects who have not undergone menopause or surgical sterilization, during the treatment period and during the study treatment
* Agree to abstain or use effective contraceptive methods for at least 2 months after the next administration; .Volunteer to join this study, sign informed consent, have good compliance, and be willing to cooperate with follow-up.

Exclusion Criteria:

* Inflammatory breast cancer
* Metastatic tumor
* Previous or concurrent malignant tumors, whose natural history or treatment may interfere with the safety of the research protocol.
* Active infections that require systemic treatment
* Has used any medication in this study within 14 days prior to enrollment
* Major surgery (excluding biopsy) performed within 14 days before enrollment

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2032-06-30 (Estimated)

PRIMARY OUTCOMES:
5-year EFS | 60 weeks
  5 years event-free survival after neoadjuvant chemoradiotherapy

SECONDARY OUTCOMES:
b-pCR | 18 weeks
  Whether combined neoadjuvant chemoradiotherapy can improve breast pathological complete response rate (bpCR: ypT0)
OS | 60 weeks
  overall survival after completing of neoadjuvant chemoradiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: XUCHEN CAO, MD, Principal Investigator — TianJin Medical University Cancer Institute and Hospitall
Locations (1):
- Tianjin medical university cancer institute and hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: Yes
Patient baseline information, patient safety information
Supporting Information: Study Protocol
Time Frame: March 30, 2027
Access Criteria: Medical scholars in the world